CLINICAL TRIAL: NCT03333070
Title: The Use of Lactobacillus Reuteri in Functional Constipation in Children: A Double Blind Randomized Control Trial
Brief Title: The Use of Lactobacillus Reuteri in Functional Constipation in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI was ended her work in the hospital and no replacement was found.
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Sarit Peleg, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0042-17-EMC
Record Dates: First submitted 2017-10-10; First posted 2017-11-06 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): 25 consecutive children diagnosed with functional constipation will be treated with full dose PEG (Polyethylene glycol 3350) treatment (dose of ~1g/kg/day) for 12 weeks.
  After 12 weeks of treatment they will be randomized: treated arm will receive probiotic containing Lactobacillus reuteri for 12 weeks while tapering the PEG dose Dose of 5 drops per day for 48 weeks
  Interventions: Dietary Supplement: probiotic - Lactobacillus reuteri
- Placebo Arm (Placebo Comparator): 25 consecutive children diagnosed with functional constipation will be treated with full dose PEG (Polyethylene glycol 3350) treatment (dose of ~1g/kg/day) for 12 weeks.
  After 12 weeks of treatment they will be randomized: control arm will receive placebo for 12 weeks while tapering the PEG dose Dose of 5 drops per day for 48 weeks
  Interventions: Other: placebo - with no active ingredient

INTERVENTIONS:
Dietary Supplement: probiotic - Lactobacillus reuteri — The treated arm will receive 5 drops per day for 48 weeks
  Arms: Treatment Arm
Other: placebo - with no active ingredient — The control arm will receive 5 drops per day for 48 weeks
  Arms: Placebo Arm

SUMMARY:
Functional constipation (FC) is a common condition in childhood, with an estimated prevalence of 0.7% to 29%.The diagnosis and treatment of FC can be difficult tasks, and children are often referred to specialist services causing treatment to become expensive and time-consuming.The standard treatment based on osmotic laxatives (mainly PEG). The recovery rate is 50% to 60% after 1 year of treatment, with 50% of the children having relapse within 5 years. Studies in adults have established the effectiveness of some lactic acid bacteria in the treatment of chronic constipation.

DETAILED DESCRIPTION:
Functional constipation (FC) is a common condition in childhood, with an estimated prevalence of 0.7% to 29%.The diagnosis and treatment of FC can be difficult tasks, and children are often referred to specialist services causing treatment to become expensive and time-consuming.The standard treatment based on osmotic laxatives (mainly PEG). The recovery rate is 50% to 60% after 1 year of treatment, with 50% of the children having relapse within 5 years. Studies in adults have established the effectiveness of some lactic acid bacteria in the treatment of chronic constipation.However, it is unclear whether similar effects occur in children. Lactobacilli and Bifidobacteria are the most studied species showing a high safety profile. Both are able to promote colonic peristalsis which could be beneficial for the treatment of constipation .Even though traditional treatment is well established and safe, high proportion of children need prolonged treatment for several months or even years. For many parents there is a concern regarding prolonged treatment with PEG .Lactobacilli, bifidobacteria and FOS (fructooligosaccharide) increase stool frequency and decrease consistency in healthy adults and therefore could prevent recurrence of constipation after PEG withdrawal .The principle investigator hypothesize that treatment with probiotics adjunct to PEG and several months thereafter could decrease the proportion of children needed permanent or prolonged treatment (>12 months) with PEG.

The importance of the study and its practical benefits:

Treatment with PEG for FC is well established and is considered safe. Despite that, a high proportion of children need prolonged treatment for several months or even years. For many parents there is a concern regarding prolonged treatment with PEG. Previous studies did not demonstrate efficacy of treatment with probiotics or prebiotics in FC. Neither of these studies assessed effectiveness probiotics/prebiotic products as adjunct to the traditional treatment (PEG) of FC in shortening its period.

A recently published studies including from Israel, demonstrated efficacy of Lactobacillus reuteri in irritable bowel syndrome, infantile colic and functional abdominal pain .Therefore, demonstration of positive effect of treatment with probiotic product in FC, could imply for potential use of this product in other functional gastrointestinal disorders among children.

ELIGIBILITY:
Inclusion Criteria:

* Age 0.5 - 15 years
* Diagnosis of functional constipation according to Rome IV criteria

Exclusion Criteria:

* Children with chronic diseases which could cause constipation: Celiac disease, food allergy, Hypothyroidism, Inflammatory Bowel Disease, electrolytes disturbances, Cystic fibrosis, Hirschsprung disease, Neuropathic conditions (Spinal cord trauma, Neurofibromatosis, Tethered cord) or intestinal pseudo-obstruction.
* Prematurity (< 34 weeks)
* S/P intestinal surgery
* Children treated with medications associated with constipation.
* Existing malignancy
* Primary or secondary immunodeficiency

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
The prevalence of constipation recurrence | This measure will be assessed at weeks 24.
  according to Rome IV criteria
The prevalence of constipation recurrence | This measure will be assessed at weeks 60.
  according to Rome IV criteria
failure of maintaining normal bowel movements without PEG and the need to resume PEG treatment | This measure will be assessed at weeks 24.
  according to Rome IV criteria
failure of maintaining normal bowel movements without PEG and the need to resume PEG treatment | This measure will be assessed at weeks 60.
  according to Rome IV criteria

SECONDARY OUTCOMES:
The number of bowel movements per week | This measure will be assessed at baseline and at 24, 36, 48 and 60 weeks after enrolment
  The investigator will collect the information during the following visits from the patient
The number of episodes of fecal incontinence per week | This measure will be assessed at baseline and at 24, 36, 48 and 60 weeks after enrolment
  The investigator will collect the information during the following visits from the patient
The stool consistency in patients without PEG treatment | This measure will be assessed at baseline and at 24, 36, 48 and 60 weeks after enrolment
  The investigator will collect the information during the following visits from the patient

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Peleg, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek medical center, Afula, Israel